CLINICAL TRIAL: NCT03841357
Title: An Open Label, Multi-Center, Phase 3 Efficacy Study of Sub-Q Abatacept in Preventing Extension of Oligoarticular Juvenile Idiopathic Arthritis JIA (Limit-JIA)
Brief Title: Preventing Extension of Oligoarticular Juvenile Idiopathic Arthritis JIA (Limit-JIA)
Acronym: Limit-JIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100523
Record Dates: First submitted 2019-01-30; First posted 2019-02-15 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Polyarthritis; abatacept; uveitis; prevention
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis; Uveitis | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Abatacept and Usual Care (Part I) (Experimental): Weekly abatacept injection at standard dosing for weight plus usual care with steroid joint injection and non-steroidal anti-inflammatory drugs per the discretion of the treating provider.
  Interventions: Drug: Abatacept Injection; Other: Usual Care
- Active Comparator: Usual Care (Part I) (Active Comparator): Usual care includes steroid joint injections and treatment with non-steroidal anti-inflammatory drugs at the discretion of the treating provider.
  Interventions: Other: Usual Care
- Abatacept and Usual Care (Part II) (Experimental): Weekly abatacept injection at standard dosing for weight plus usual care with steroid joint injection and non-steroidal anti-inflammatory drugs per the discretion of the treating provider.
  Interventions: Drug: Abatacept Injection; Other: Usual Care
- Active Comparator: Usual Care (Part II) (Active Comparator): Usual care includes steroid joint injections and treatment with non-steroidal anti-inflammatory drugs at the discretion of the treating provider.
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: Abatacept Injection — Supplied as a weekly injection via a pre-filled syringe
  Other Names: Orencia
  Arms: Abatacept and Usual Care (Part I); Abatacept and Usual Care (Part II)
Other: Usual Care — Usual care will be defined by the clinical management team but includes steroid joint injections and non- steroidal anti-inflammatory drugs

SUMMARY:
This is a research study to test whether a once-weekly injection of abatacept will prevent the progression of Juvenile Idiopathic Arthritis (JIA) to a more severe form. To evaluate the effectiveness of a 24-week course of treatment with abatacept plus usual care versus usual care to prevent polyarthritis (≥5 joints), uveitis, or treatment with other systemic medication within 18 months of randomization in children with recent-onset limited JIA.

DETAILED DESCRIPTION:
Part I enrolled participants into a randomized open-label multicenter trial with a planned sample size of 306 JIA participants recruited from CARRA Registry sites. Participants were randomly allocated (1:1) to receive 24 weeks of abatacept plus usual care or usual care alone. Upon completion of 24 weeks of randomized treatment, each participant was to receive usual care and undergo follow-up for assessment of outcomes for an additional 12 months. Planned duration of the study for each participant was 18 months. Due to slow accrual and apparent loss of equipoise, enrollment into Part I was discontinued. Part I participants continued follow-up as planned.

Part II is a non-randomized continuation of LIMIT-JIA with planned enrollment of 89 to reach 80 evaluable participants receiving to the abatacept arm. Participants will now receive 24 doses of abatacept plus usual care. Upon completion of 24 doses of treatment, each participant will receive usual care and undergo follow-up for assessment of outcomes for an additional 6 months. Planned duration of the study for each participant is 12 months. Part II will assess the efficacy of abatacept in prevention of disease extension by comparison of outcomes between participants enrolled in the abatacept arm and CARRA Registry patients who would have met major eligibility criteria for LIMIT-JIA.

ELIGIBILITY:
To be eligible for this trial, participants must meet all of the following criteria in order to be include in the study:

1. Age ≥ 2 years old and ≤16.5 years old
2. Clinical diagnosis of JIA by a pediatric rheumatologist within the past 6 months
3. Arthritis affecting ≤4 joints between disease onset and enrollment
4. Enrollment in the CARRA Registry
5. Participants of childbearing potential must agree to remain abstinent or agree to use an effective and medically acceptable form of birth control from the time of written or verbal assent to at least 66 days after taking the last dose of study drug.
6. Weight ≥50 kg (Canadian Sites only) ¹ Enrollment is defined as having signed consent to participate in the Limit-JIA study.

The presence of any of the following will exclude a study participant from inclusion in the study:

1. 1. Systemic JIA as defined by 2004 ILAR criteria1
2. Sacroiliitis (clinical or radiographic)
3. Inflammatory bowel disease (IBD)
4. History of psoriasis or currently active psoriasis
5. History of uveitis or currently active uveitis
6. Prior treatment with systemic medication(s) for JIA (e.g. one or more of the following: DMARD or biologic medication)
7. Current or previous (within 30 days of enrollment) treatment with systemic glucocorticoids (A short course of oral prednisone [≤ 14 days] is allowed)
8. History of active or chronic liver disease
9. Chronic or acute renal disorder
10. AST (SGOT), ALT (SGPT) or BUN >2 x ULN (upper limit of normal) or creatinine >1.5 mg/dL or any other laboratory abnormality considered by the examining physician to be clinically significant within 2 months of the enrollment visit
11. Presence of any medical or psychological condition or laboratory result which would make the participant, in the opinion of the investigator, unsuitable for the study
12. Participation in another concurrent clinical interventional study within 30 days of enrollment
13. Known positive human immunodeficiency virus (HIV)
14. Received a live virus vaccine within 1 month of the baseline visit
15. Current or prior positive Purified Protein Derivative (PPD) test or Quantiferon Gold TB
16. Pregnant, breast feeding, or planned breast feeding during the study duration
17. Planned transfer to non-participating pediatric rheumatology center or adult rheumatologist in the next 12 months
18. Active malignancy of any type or history of malignancy
19. Chronic or active infection or any major episode of infection requiring hospitalization or treatment with intravenous (IV) antibiotics within 30 days or oral antibiotics within 14 days prior to screening
20. Primary language other than English or Spanish
21. Positive for Hepatitis B surface antigen or core antibody
22. <10 Kg in weight
23. If a potential subject has symptoms consistent with COVID-19 and/or known COVID-19 exposure at screening, it is recommended that the site follow CDC guidance regarding testing and quarantine requirements. The subject can be re-screened when there is no longer concern for active infection. A subject with a positive COVID -19 test may be re-screened.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Schanberg, MD, Principal Investigator — Duke University; Eveline Wu, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (19):
- United States (19):
  - University of California at San Francisco Medical Center, San Francisco, California
  - The Children's Hospital Colorado, Aurora, Colorado
  - Shands at the University of Florida, Gainesville, Florida
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - University of Iowa Hospitals of Clinics, Iowa City, Iowa
  - University of Louisville School of Medicine/ Norton Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota; Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Children's Hospital at Montefiore/ Albert Einstein University Hospital, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - MetroHealth System, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Usual Care (Part II) participants were historical controls used for analysis and not considered enrolled.
Period: Overall Study
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II)
Started | 20 | 20 | 81 | 662
Completed | 20 | 20 | 80 | 662
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II) | Total
Number analyzed (Participants) | 20 | 20 | 81 | 662 | 783
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.90 (4.60) | 6.10 (4.40) | 7.60 (4.20) | 7.60 (4.35) | 7.57 (4.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 55 | 438 | 516
  Male | 9 | 8 | 26 | 224 | 267
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 16 | 66 | 87
  Not Hispanic or Latino | 17 | 18 | 65 | 594 | 694
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 2
  Asian | 0 | 1 | 0 | 17 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 2 | 2
  Black or African American | 1 | 1 | 2 | 28 | 32
  White | 14 | 13 | 56 | 486 | 569
  More than one race | 3 | 2 | 10 | 55 | 70
  Unknown or Not Reported | 2 | 3 | 13 | 72 | 90
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 81 | 662 | 783

OUTCOME MEASURES:

1. Primary Outcome: Composite of All Primary Endpoints
Description: Any of the following from randomization to day 410: polyarthritis [>=5 cumulative active joint count], uveitis, initiation of systemic glucocorticoids (IV or PO), DMARDs or biologics.
Time Frame: From randomization to day 410
Population: Modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Groups:
- Abatacept and Usual Care (Part I); Abatacept and Usual Care (Part II); Abatacept and Usual Care (Pooled Part I and Part II): Weekly abatacept injection at standard dosing for weight plus usual care with steroid joint injection and non-steroidal anti-inflammatory drugs per the discretion of the treating provider.
  Abatacept Injection: Supplied as a weekly injection via a pre-filled syringe
  Usual Care: Usual care will be defined by the clinical management team but includes steroid joint injections and non-steroidal anti-inflammatory drugs
- Active Comparator: Usual Care (Part I); Active Comparator: Usual Care (Part II); Active Comparator: Usual Care (Pooled Part I and Part II): Usual care includes steroid joint injections and treatment with non-steroidal anti-inflammatory drugs at the discretion of the treating provider.
  Usual Care: Usual care will be defined by the clinical management team but includes steroid joint injections and non-steroidal anti-inflammatory drugs
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II) | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 20 | 20 | 76 | 596 | 96 | 616
Participants | 13 | 14 | 41 | 245 | 54 | 259
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Part I) vs Active Comparator: Usual Care (Part I); The null hypothesis was the proportions of the patients with composite of primary endpoints were the same between two groups; Test type: Superiority; p = 0.7357, Cochran-Mantel-Haenszel; Relative Risk = 0.929, 95% CI 2-sided [0.603 to 1.429], Standard Error of Mean 0.220
Statistical Analysis 2: Comparison: Abatacept and Usual Care (Part II) vs Active Comparator: Usual Care (Part II); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Relative Risk = 1.16, 95% CI 2-sided [0.90 to 1.48]
Statistical Analysis 3: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Relative Risk = 1.19, 95% CI 2-sided [0.93 to 1.51]

2. Primary Outcome: Number of Participants With Polyarthritis
Description: Polyarthritis is defined as >=5 cumulative active joint count.
Time Frame: From randomization to day 592
Population: Modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II) | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 20 | 20 | 76 | 596 | 96 | 616
Participants | 8 | 6 | 14 | 49 | 22 | 55
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Part I) vs Active Comparator: Usual Care (Part I); The null hypothesis was the proportions of the patients with this primary endpoint were the same between two groups; Test type: Superiority; p = 0.507, Cochran-Mantel-Haenszel; Relative Risk = 1.333, 95% CI 2-sided [0.565 to 3.145], Standard Error of Mean 0.438
Statistical Analysis 2: Comparison: Abatacept and Usual Care (Part II) vs Active Comparator: Usual Care (Part II); The null hypothesis was the proportions of the patients with this primary endpoint were the same between two groups; Test type: Superiority; Relative Risk = 1.00, 95% CI 2-sided [0.38 to 2.59]
Statistical Analysis 3: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); The null hypothesis was the proportions of the patients with this primary endpoint were the same between two groups; Test type: Superiority; Relative Risk = 1.35, 95% CI 2-sided [0.77 to 2.37]

3. Primary Outcome: Number of Participants With Uveitis
Time Frame: From randomization to day 410
Population: Modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II) | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 20 | 20 | 76 | 596 | 96 | 616
Participants | 1 | 0 | 4 | 31 | 5 | 31
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Part II) vs Active Comparator: Usual Care (Part II); The null hypothesis was the proportions of the patients with this primary endpoint were the same between two groups; Test type: Superiority; Relative Risk = 0.97, 95% CI 2-sided [0.32 to 2.92]
Statistical Analysis 2: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); The null hypothesis was the proportions of the patients with this primary endpoint were the same between two groups; Test type: Superiority; Relative Risk = 1.00, 95% CI 2-sided [0.29 to 3.38]

4. Primary Outcome: Number of Participants With Systemic Medications
Description: Systemic glucocorticoids, Disease-Modifying Antirheumatic Drugs (DMARDs) or biologics.
Time Frame: From randomization day 410
Population: Modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II) | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 20 | 20 | 76 | 596 | 96 | 616
Participants | 11 | 14 | 41 | 229 | 52 | 243
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Part I) vs Active Comparator: Usual Care (Part I); The null hypothesis was the proportions of the patients with this primary endpoint were the same between two groups; Test type: Superiority; p = 0.327, Cochran-Mantel-Haenszel; Relative Risk = 0.786, 95% CI 2-sided [0.482 to 1.282], Standard Error of Mean 0.250
Statistical Analysis 2: Comparison: Abatacept and Usual Care (Part II) vs Active Comparator: Usual Care (Part II); The null hypothesis was the proportions of the patients with this primary endpoint were the same between two groups; Test type: Superiority; Relative Risk = 1.06, 95% CI 2-sided [0.53 to 2.09]
Statistical Analysis 3: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); The null hypothesis was the proportions of the patients with this primary endpoint were the same between two groups; Test type: Superiority; Relative Risk = 1.19, 95% CI 2-sided [0.90 to 1.59]

5. Secondary Outcome: Number of Participants With Clinically Inactive Disease or Remission
Description: Clinical Inactive disease at any visit is a composite outcome consisting of all of: No active joints (Current Active Joint Count=0), No uveitis (Uveitis=No or not reported), Normal ESR (if obtained) (N/D or ESR≤ ULN or unrelated to JIA if >ULN), Normal CRP (if obtained) (N/D or CRP≤ ULN or unrelated to JIA if >ULN), AM stiffness duration=None or ≤ 15 minutes, Physician Global score=0.
Time Frame: From baseline up to 12 months
Population: Intent-to-treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II) | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 20 | 20 | 80 | 662 | 100 | 682
Participants | 8 | 3 | 36 | 246 | 48 | 264
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Part II) vs Active Comparator: Usual Care (Part II); The null hypothesis was the proportions of the patients with this primary endpoint were the same between two groups; Test type: Superiority; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.05 to 2.13]
Statistical Analysis 2: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); The null hypothesis was the proportions of the patients with this primary endpoint were the same between two groups; Test type: Superiority; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.08 to 2.04]

6. Secondary Outcome: Number of Participants With Disease Extension
Description: Disease extension defined as development of polyarthritis or uveitis.
Time Frame: From baseline up to 12 months
Population: Intent-to-treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II) | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 20 | 20 | 80 | 662 | 100 | 682
Participants | 7 | 6 | 11 | 67 | 18 | 73
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Part II) vs Active Comparator: Usual Care (Part II); Test type: Superiority; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.53 to 2.35]
Statistical Analysis 2: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); Test type: Superiority; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.76 to 2.24]

7. Secondary Outcome: Number of New Active Joints Per Participant
Description: Total number of joints that were not active prior to or at baseline, and became active after randomization.
Time Frame: From baseline up to 12 months
Population: Intent-to-treat (ITT) population.
Measure: Mean (Standard Error); unit: joints
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II) | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 20 | 20 | 80 | 662 | 100 | 682
joints | 1.40 (1.67) | 1.50 (1.57) | 0.70 (1.69) | 0.40 (1.43) | 0.80 (1.70) | 0.50 (1.44)
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Part II) vs Active Comparator: Usual Care (Part II); Test type: Superiority; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.48 to 2.19], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); Test type: Superiority; Risk Ratio (RR) = 1.29, 95% CI 2-sided [0.74 to 2.24], Standard Error of Mean 0.36

8. Secondary Outcome: Number of Intra-articular Glucocorticoid Joint Injections Per Participant
Description: Intra-articular glucocorticoid joint injections are reported in the CARRA Registry CRF at each Limit-JIA or CARRA Registry visit.
Time Frame: From baseline up to 12 months
Population: Intent-to-treat (ITT) population.
Measure: Mean (Standard Error); unit: injections
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II) | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 20 | 20 | 80 | 662 | 100 | 682
injections | 0.90 (1.17) | 1.80 (2.61) | 0.40 (1.31) | 0.40 (0.85) | 0.50 (1.29) | 0.40 (0.97)
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Part II) vs Active Comparator: Usual Care (Part II); Test type: Superiority; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.49 to 2.17], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); Test type: Superiority; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.64 to 1.89], Standard Error of Mean 0.30

9. Secondary Outcome: PROMIS (Patient-Reported Outcomes Measurement Information System) Pediatric Pain Interference
Description: PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS scores are T-scores and have a mean of 50 and standard deviation of 10.
Time Frame: 6 months and 12 months
Population: Pooled intent-to-treat (ITT) population with data collected at each timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 44 | 234
score on a scale
  6 months: number analyzed (Participants) | 37 | 234
  6 months | 49.00 (9.81) | 50.90 (8.72)
  12 months: number analyzed (Participants) | 44 | 190
  12 months | 46.90 (9.87) | 49.60 (9.91)
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); Test type: Superiority; p = 0.005, Mixed Models Analysis; Difference in Least Square Means = -1.23, 95% CI 2-sided [-2.09 to -0.38], Standard Error of Mean 0.44

10. Secondary Outcome: PROMIS (Patient-Reported Outcomes Measurement Information System) Pediatric Fatigue
Description: as for outcome 9
Time Frame: 6 months and 12 months
Population: Pooled intent-to-treat (ITT) population with data collected at each timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 65 | 10
score on a scale
  6 months | 39.60 (8.94) | 43.50 (13.85)
  12 months: number analyzed (Participants) | 56 | 10
  12 months | 39.80 (9.12) | 47.10 (16.85)
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); Test type: Superiority; p = 0.174, Mixed Models Analysis; Difference in Least Square Means = -4.85, 95% CI 2-sided [-11.86 to 2.16], Standard Error of Mean 3.58

11. Secondary Outcome: PROMIS (Patient-Reported Outcomes Measurement Information System) Upper Extremity Function
Description: as for outcome 9
Time Frame: 6 months and 12 months
Population: Pooled intent-to-treat (ITT) population with data collected at each timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 59 | 221
score on a scale
  6 months | 44.30 (12.73) | 42.20 (12.61)
  12 months: number analyzed (Participants) | 46 | 184
  12 months | 44.10 (11.87) | 42.30 (12.82)
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); Test type: Superiority; p = 0.012, Mixed Models Analysis; Difference in Least Square Means = 1.57, 95% CI 2-sided [0.35 to 2.80], Standard Error of Mean 0.63

12. Secondary Outcome: PROMIS (Patient-Reported Outcomes Measurement Information System) Mobility
Description: as for outcome 9
Time Frame: 6 months and 12 months
Population: Pooled intent-to-treat (ITT) population with data collected at each timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 76 | 365
score on a scale
  6 months | 51.00 (9.28) | 49.20 (8.77)
  12 months: number analyzed (Participants) | 74 | 320
  12 months | 50.30 (8.38) | 50.70 (8.79)
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in Least Square Means = 1.53, 95% CI 2-sided [0.69 to 2.37], Standard Error of Mean 0.43

13. Secondary Outcome: PROMIS (Patient-Reported Outcomes Measurement Information System) Anxiety
Description: as for outcome 9
Time Frame: 6 months
Population: Pooled intent-to-treat (ITT) population with data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 73 | 12
score on a scale | 40.60 (8.23) | 43.60 (10.87)

14. Secondary Outcome: PROMIS (Patient-Reported Outcomes Measurement Information System) Depression
Description: as for outcome 9
Time Frame: 6 months
Population: Pooled intent-to-treat (ITT) population with data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 74 | 12
score on a scale | 40.00 (7.18) | 43.30 (9.39)

15. Secondary Outcome: PROMIS (Patient-Reported Outcomes Measurement Information System) Global Health
Description: as for outcome 9
Time Frame: 6 months and 12 months
Population: Pooled intent-to-treat (ITT) population with data collected at each timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 77 | 399
score on a scale
  6 months | 42.50 (6.51) | 42.10 (4.89)
  12 months: number analyzed (Participants) | 74 | 339
  12 months | 43.00 (5.84) | 42.70 (5.41)
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); Test type: Superiority; p = 0.002, Mixed Models Analysis; Difference in Least Square Means = 0.74, 95% CI 2-sided [0.28 to 1.20], Standard Error of Mean 0.24

16. Secondary Outcome: Juvenile Arthritis Disease Activity Score (JADAS)
Description: The JADAS (Juvenile Arthritis Disease Activity Score) is a composite tool used to assess disease activity in children with Juvenile Idiopathic Arthritis (JIA). The total score ranges from 0 to 40, where a higher score indicates a more severe level of disease activity.
Time Frame: 6 months and 12 months
Population: Pooled intent-to-treat (ITT) population with data collected at each timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Abatacept and Usual Care (Pooled Part I and Part II) | Active Comparator: Usual Care (Pooled Part I and Part II)
Number analyzed (Participants) | 89 | 457
score on a scale
  6 months | 2.60 (3.23) | 3.00 (3.29)
  12 months: number analyzed (Participants) | 87 | 408
  12 months | 2.50 (3.15) | 2.60 (3.06)
Statistical Analysis 1: Comparison: Abatacept and Usual Care (Pooled Part I and Part II) vs Active Comparator: Usual Care (Pooled Part I and Part II); Test type: Superiority; p < 0.001, Mixed Models Analysis; Difference in Least Square Means = -0.55, 95% CI 2-sided [-0.84 to -0.26], Standard Error of Mean 0.15

17. Other Pre Specified Outcome: Elapsed Time From Randomization to Primary Endpoint
Description: Time from enrollment to the earliest of the following: Date of visit when polyarthritis is first noted, Date of eye exam when Uveitis is first reported, Date of first reported use of systemic DMARDs and/or Biologics, including systemic glucocorticoids (IV or PO).
Time Frame: From randomization up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Only Events of Special Interest (ESIs), serious and non-serious, and SAEs were collected for this study.
Arm/Group | Abatacept and Usual Care (Part I) | Active Comparator: Usual Care (Part I) | Abatacept and Usual Care (Part II) | Active Comparator: Usual Care (Part II)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/80 | 0/662
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 3/80 | 0/662
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/80 | 0/662
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept and Usual Care (Part I) (N=20) | Active Comparator: Usual Care (Part I) (N=20) | Abatacept and Usual Care (Part II) (N=80) | Active Comparator: Usual Care (Part II) (N=662)
COVID-19 infection (Infections and infestations) | 1 | 0 | 0 | 0
Malignancy, B-cell acute lymphoblastic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Blood streaked emesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Infection treated with IV anti-infectives (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT03841357/Prot_SAP_000.pdf